CLINICAL TRIAL: NCT00977678
Title: Drop in Gastroscopy - Experience After 9 Months
Status: Completed | Type: Observational
Sponsor: Norwegian Department of Health and Social Affairs (Other Government)
Responsible Party: Gert Huppertz-Hauss, Telemark Hospital, N-3710 Skien, Norway
Other Study IDs: STHF-1
Record Dates: First submitted 2009-05-15; First posted 2009-09-16 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Diseases; Peptic Ulcer; Stomach Diseases
Keywords: open access gastroscopy
MeSH Terms: conditions — Esophageal Diseases; Peptic Ulcer; Stomach Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Open access gastroscopy: Patients referred to open access gastroscopy
  Interventions: Other: open access gastroscopy
- Conventional outpatient gastroscopy: Gastroscopy after preceding appointment
  Interventions: Other: Gastroscopy by appointment

INTERVENTIONS:
Other: open access gastroscopy — access to gastroscopy without preceding appointment
  Groups: Open access gastroscopy
Other: Gastroscopy by appointment — Gastroscopy after preceding appointment in a conventional outpatient clinic
  Groups: Conventional outpatient gastroscopy

SUMMARY:
The capacity for endoscopical procedures in the Norwegian health system is low in comparison to demands from patients and family practitioners.

The studies aim is to evaluate the acceptance of a new concept: an open access gastroscopy clinic where patients can attend without a preceding appointment.

The investigators wish to evaluate:

1. Patient´s satisfaction.
2. General practitioner´s satisfaction.
3. Acceptance by the staff of the clinic.

DETAILED DESCRIPTION:
The fact that access to specialized norwegian health care is characterized by a mismatch between system´s capacity and patient´s and refering physician´s demands, leads to delay of diagnostic investigations such as for example gastroscopies. Patients referred to gastroscopies have to wait 4 to 12 weeks to get an appointment. Consequence might be a delay in diagnosing of significant diseases such as ulcers or even malignancies. In addition the general practitioner is frequently forced to start a therapy by suspicion, and the patient has in numerable cases to stay off work.

In September 2008, the investigators started an open-access gastroscopy outpatient clinic, which allows the family practitioners in a defined area of the Telemark county to refer their patients to a gastroscopy without a preceding appointment. Patients from the other parts of the county and those, who need special service as i.e. interpreter, endocarditis prophylaxis etc. are referred conventionally and need an appointment.

Aim of the study is to evaluate the acceptance of both forms of outpatient clinics by both patients and general practitioners. In addition to that, the investigators will evaluate the acceptance of the open access clinic by the staff. Of special concern is the fear, that easier access might lead to a number of unnecessary procedures.

All patients from open access clinic and from the conventional clinic are asked to fill in a questionaire without any kind of personal identifying data such as name, age, date of the procedure etc., but with questions about their satisfaction with the procedure, the time from their first contact with their family practitioner to the procedure, the information prior and after the procedure. They will be asked if they did consume drugs against "ulcer-disease" or not.

In addition the referring practitioners are asked to fill in a questionnaire about their acceptance of the open access clinic, and to give the investigators some ideas about advantages and disadvantages from their point of view.

The staff is asked to give their experience especially according to the not calculable number of patients that attend to the clinic each day.

If the present study shows high acceptance of the open-access-offer by patients and health workers, the plan is to extend it to other patient groups and to perform studies to investigate the effects on the grade of diseases at the time of diagnosis and possible consequences for treatment and health economy.

ELIGIBILITY:
Inclusion Criteria:

* all patients from 18 years of age.

Exclusion Criteria:

* age < 18,
* inability or unwillingness to cooperate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current patients referred to our outpatient gastroscopy clinic
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Patient´s satisfaction | Day of the Gastrocopy

SECONDARY OUTCOMES:
General practitioner´satisfaction | One month after enrollment of patients

CONTACTS AND LOCATIONS:
Overall Officials: Gert Huppertz-Hauss, MD, Principal Investigator — Telemark Hospital, Department of internal medicin, Skien, Norway
Locations (1):
- Department of Gastroenterology, Skien, Telemark, Norway